CLINICAL TRIAL: NCT03065192
Title: An Open-label Safety and Efficacy Study of VY-AADC01 Administered by MRI-Guided Convective Infusion Using a Posterior Trajectory Into the Putamen of Participants With Parkinson's Disease With Fluctuating Responses to Levodopa
Brief Title: Safety and Efficacy Study of VY-AADC01 for Advanced Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Voyager Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1102
Record Dates: First submitted 2017-02-10; First posted 2017-02-27 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Parkinson's Disease; Parkinson's Disease; Basal Ganglia Disease; Brain Diseases; Central Nervous System Diseases; Movement Disorders; Nervous System Diseases; Neurodegenerative Diseases; Parkinsonian Disorders
Keywords: Gene Therapy; PD; Parkinson's Disease; Aromatic L- Amino Acid Decarboxylase; AADC; AAV2-AADC; AAV2; Viral Vector; Gene Transfer; MRI; PET; VY-AADC01
MeSH Terms: conditions — Parkinson Disease; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Movement Disorders; Nervous System Diseases; Neurodegenerative Diseases; Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VY-AADC01 Single Dose (Experimental): 9.4 x 10^12 vector genomes of VY-AADC01
  Interventions: Drug: VY-AADC01

INTERVENTIONS:
Drug: VY-AADC01 — Single dose, neurosurgically infused, bilaterally into the striatum.

SUMMARY:
Safety and efficacy of AADC gene transfer in participants with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder involving loss of dopamine producing neurons located in the striatum. Levodopa is the primary treatment used to treat Parkinson's disease, which converts to dopamine by the enzyme (protein) Aromatic L-Amino Acid Decarboxylase (AADC). As PD progresses, the amount of AADC levels in the brain decreases, and in turn, reduces the amount of dopamine that is produced with each dose of levodopa.

The primary objective of this study is to evaluate the safety of increasing AADC levels, via gene delivery. The investigational drug, termed VY-AADC-01, will be injected directly into the striatum during a neurosurgical procedure that is performed with real-time MRI imaging to monitor delivery.

Participants will continue to take their Parkinson medications, including levodopa while participating in this study.

The safety and potential clinical responses to VY-AADC-01 will be assessed by repeated clinical evaluations of Parkinson's disease, treatment review phone calls, cognitive tests, laboratory blood tests, patient reported outcomes scales, patient diaries, collection of adverse events, and neuro-imaging. Clinical evaluations will be performed over a 3 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic PD.
* Adequate duration of levodopa therapy.
* Disease duration of at least 5 years or more.
* Modified Hoehn & Yahr Staging with at least 2.5 hours or more in the OFF state.
* Candidate for surgical intervention because of disabling motor complications.
* UPDRS Part III (total score) of at least 25 in the OFF state.
* Unequivocal responsiveness to dopaminergic therapy.
* Stable Parkinson's symptoms and medications for at least 4 weeks prior to screening evaluation.
* Ability to comprehend and sign the informed consent.
* Normal laboratory values prior to surgery.
* Medically and mentally capable of undergoing and complying with the surgical procedure and protocol requirements.
* Ability to travel to study visits alone or able to designate a caregiver.
* Subject agrees to defer any neurological surgery, including deep brain stimulation, until after completing the 12 month study visit (unless recommended by study neurologist).
* Approved by the Eligibility Review Committee.

Exclusion Criteria:

* Atypical or secondary parkinsonism, including but not limited to symptoms believed to be due to trauma, brain tumor, infection, cerebrovascular disease, other neurological disease, or to drugs, chemicals, or toxins.
* Presence of dementia as defined by a Mattis Dementia Rating Scale - Second Edition (MDRS-2) score of less than 130 at screening.
* Presence or history of psychosis, with the exception of mild, benign hallucinations believed in the judgment of the Investigator to be related to Parkinson's medications.
* Presence of severe depression, as indicated by a BDI-II score greater than 28, or a history of a major affective disorder within 5 years of screening evaluation.
* Active suicidal ideation or suicide attempt within 5 years of screening evaluation.
* History of substance abuse within 2 years of screening evaluation.
* Brain imaging abnormalities in the striatum or other regions that would substantially increase risk of surgery.
* Contraindication to MRI and/or gadoteridol.
* Coagulopathy or inability to temporarily stop any anticoagulation or antiplatelet therapy prior to surgery.
* Prior brain surgery including lesioning procedures, deep brain stimulation, infusion therapies or any other brain surgery.
* Prior gene transfer.
* History of stroke, poorly controlled or significant cardiovascular disease, diabetes, or any other acute or chronic medical condition.
* History of malignancy other than treated carcinoma in situ within 3 years of screening evaluation.
* Clinically apparent or laboratory-detected infection.
* Prior or current treatment with any investigational agent within 2 months of screening evaluation.
* Inability to comply with the procedures of the protocol, including completion of paper Parkinson's disease diaries, frequent and prolonged study visits including off medication visits, and travel.
* Chronic immunosuppressive therapy, including chronic steroids, immunotherapy, cytotoxic therapy, and chemotherapy.
* Any serious medical condition or abnormal finding on physical examination or laboratory investigation that would substantially increase the risks of the study procedures.
* Any medical condition that is likely to lead to disability during the course of the study and interfere with or confound study assessments.
* Pregnant and lactating women.
* Male or female with reproductive capacity who is unwilling to use barrier contraception for 6 months after surgery.
* Plans to receive any vaccination within 30 days of surgery.
* Any factors, medical or social, which would likely cause the participant to be unable to follow the study protocol, including geographical inaccessibility.
* Ongoing treatments including neuroleptic medications, apomorphine, or levodopa infusion therapy (Duopa®).
* Plans to participate in any other therapeutic intervention study within 12 months after surgery.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Grading of adverse Events/Serious Adverse Events (AE's/SAE's) | Baseline to 3 Years After Gene Transfer
  Grading will be assessed using NCI CTCAE, version 4.03.
Magnetic Resonance Imaging (MRI) | Baseline to 3 Years After Gene Transfer
  Safety of VY-AADC01 will be assessed by any clinically significant abnormalities on MRI scans as compared to Baseline.
Routine physical examinations | Baseline to 3 Years After Gene Transfer
  Safety of VY-AADC01 will be assessed by routine physical examinations.
Routine clinical laboratory analysis | Baseline to 3 Years After Gene Transfer
  Safety of VY-AADC01 will be assessed by routine clinical laboratory analysis.
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) results | Baseline to 3 Years After Gene Transfer
  C-SSRS is a standardized suicidal rating system.

SECONDARY OUTCOMES:
Change in Parkinson's medications | Baseline to 3 Years After Gene Transfer
  Change in Parkinson's medications compared to Baseline.
Change in motor function using Parkinson Disease Diaries | Baseline to 3 Years After Gene Transfer
  Diary used to assess changes in PD motor symptoms.
Change in motor function using a Stand-Walk-Sit Test | Baseline to 3 Years After Gene Transfer
  Standardized test used in PD studies to assess functional mobility.
Change in motor function using Modified Hoehn and Yahr Scale | Baseline to 3 Years After Gene Transfer
  Scale used to measure overall level of disability due to PD.
Change in motor function using Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline to 3 Years After Gene Transfer
  Standard assessment scale used to quantify signs and symptoms of PD.
Change in occurrence of dyskinesia using Unified Dyskinesia Rating Scale (UDysRS) | Baseline to 3 Years After Gene Transfer
  Comprehensive rating tool used to assess essential features of dyskinesia in PD.
Change in mood using Beck Depression Inventory II (BDI-II) | Baseline to 3 Years After Gene Transfer
  Self-administered measure of depression symptoms.
Change in cognitive function using Modified Cognitive Assessment (MoCA) | Baseline to 3 Years After Gene Transfer
  Rapid screening instrument for mild cognitive dysfunction.
Change in cognitive function using Mattis Dementia Rating Scale - Second Edition (MDRS-2) | Baseline to 3 Years After Gene Transfer
  Standardized neuropsychological test battery to measure dementia.
Change in compulsive behavior using the Questionnaire Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) | Baseline to 3 Years After Gene Transfer
  Rating scale to quantify the severity of a variety of compulsive disorders and behaviors.
Change in sleep quality and disturbance using the Parkinson's Disease Sleep Scale 2 (PDSS-2) | Baseline to 3 Years After Gene Transfer
  Visual analogue scale addressing 15 commonly reported symptoms associated with sleep disturbance in PD.
Change in Non-Motor System Scale (NMSS) | Baseline to 3 Years Gene Transfer
  Standard rating scale that assesses the non-motor symptoms that may be associated with PD.
Change in quality of life using Parkinson's Disease Questionnaire (PDQ39) | Baseline to 3 Years After Gene Transfer
  Validated questionnaire to measure health related quality of life in PD patients.
Change in quality of life using Schwab and England Scale | Baseline to 3 Years After Gene Transfer
  PD specific disability scale used to express the levels of independence with activities of daily living.
Change in quality of life using in Clinical Global Impression Scale (CGI) | Baseline to 3 Years After Gene Transfer
  Scale used to assess treatment response in psychiatric patients.
Change in quality of life using Patient Global Impression Scale (PGI) | Baseline to 3 Years After Gene Transfer
  Scale used to assess participants improvement in their PD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Hersch, MD, Study Director — Voyager Therapeutics, Inc.
Locations (4):
- United States (4):
  - University of California, San Francisco (UCSF), San Francisco, California
  - Emory University, Atlanta, Georgia
  - Ohio State University (OSU), Columbus, Ohio
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company Website — http://voyagertherapeutics.com/